CLINICAL TRIAL: NCT04437004
Title: Treatment of Dravet Syndrome With Fenfluramine (Expanded Access Protocol)
Acronym: Dravet
Status: Available | Type: Expanded Access
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Shaun Hussain, MD, Associate Professor, University of California, Los Angeles
Other Study IDs: ZX008-1800
Record Dates: First submitted 2020-02-21; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Fenfluramine

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Fenfluramine — The treatment plan for this Expanded Access Protocol is for patients with Dravet syndrome who do not qualify for participation in one of the ongoing ZX008 (fenfluramine hydrochloride) clinical trials.
  Other Names: Fenfluramine Hydrochloride

SUMMARY:
The purpose of this research study is to (1) provide access to fenfluramine for patients with intractable epilepsy associated with Dravet syndrome, and (2) evaluate the safety of fenfluramine.

DETAILED DESCRIPTION:
The purpose of this research study is to (1) provide access to fenfluramine for patients with intractable epilepsy associated with Dravet syndrome, and (2) evaluate the safety of fenfluramine.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of Dravet syndrome with intractable seizures despite failing all available medications for seizures.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States